CLINICAL TRIAL: NCT05790408
Title: Anterior-segment OCT (AS-OCT) and Intraoperative OCT (iOCT) for Trans- Conjunctival Needle Revision (TCNR) of Trabeculectomy Bleb
Brief Title: Anterior-segment OCT (AS-OCT) and Intraoperative OCT (iOCT) for Trans- Conjunctival Needle Revision (TCNR)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment, lack of availability of equipment, lack of availability of staff
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Angelo P Tanna, Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00213080
Record Dates: First submitted 2022-01-04; First posted 2023-03-30 (Actual); Results first posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-10

CONDITIONS: Glaucoma; Glaucoma Following Surgery
Keywords: optical coherence tomography
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- AS-OCT and iOCT (Other): This prospective study will include approximately 25 patients with open-angle glaucoma who will undergo TCNR of trabeculectomy bleb by a glaucoma specialist at Northwestern Medicine. These patients will have a history of glaucoma and failed trabeculectomy bleb (as evidenced by clinical features and elevated IOP). During routine clinic visit, the patient will undergo lit lamp grading of bleb by Indiana Bleb Appearance Grading Score (IBAGS). Subjects who agree to participate and provide written informed consent will undergo AS-OCT imaging (Spectralis OCT, Heidelberg) of the bleb. During their operation, the Zeiss Artevo digital microscope integrated with iOCT (Zeiss Artevo 800, Carl Zeiss Meditec AG), a commercially available device will be utilized to visualize and evaluate the morphology of the trabeculectomy bleb at the start and conclusion of the case.
  Interventions: Device: Digital microscope integrated with intraoperative OCT (Zeiss Artevo 800, Carl Zeiss Meditec AG); Device: Spectralis Anterior-segment OCT (AS-OCT) (Heidelberg Engineering)

INTERVENTIONS:
Device: Digital microscope integrated with intraoperative OCT (Zeiss Artevo 800, Carl Zeiss Meditec AG) — The Zeiss Artevo digital microscope integrated with iOCT (Zeiss Artevo 800, Carl Zeiss Meditec AG) is a commercially available, FDA approved device that can be utilized to visualize and evaluate the morphology of the trabeculectomy bleb during transconjunctival needle revision of trabeculectomy bleb.
Device: Spectralis Anterior-segment OCT (AS-OCT) (Heidelberg Engineering) — The Spectralis Anterior-segment OCT (AS-OCT) is a commercially available, FDA approved device that can be utilized to visualize and evaluate the morphology of the trabeculectomy bleb in the office.

SUMMARY:
Trabeculectomy is a very important and commonly performed glaucoma operation. It allows fluid from inside the eye to exit into a space called a bleb located on the surface of the eye under the upper eyelid. The formation of excessive scar tissue after surgery may cause the operation to work less well or stop working. This results in an increase in eye pressure. The use of a needle to cut the scar tissue is a commonly used procedure. This surgery is called trans-conjunctival needle revision (TCNR) of trabeculectomy bleb.

The study aims to determine if advanced optical imaging called Optical Coherence Tomography (OCT) of the scar tissue both in the office prior to surgery and during surgery in the operating room improves the success rate of the revision surgery. These devices are FDA approved and have been used extensively in ophthalmology and ocular surgery.

Ophthalmologists already used these imaging devices for this purpose as part of the standard medical care of some patients. The purpose of this study is to prospectively gather information about its use in a systematic way. Furthermore, investigators want to determine if imaging improves outcomes compared to historical controls (patients who underwent the same surgery in the past without imaging). The potential benefit of this research is that it may provide knowledge that will be of benefit to future patients with glaucoma who are undergoing this procedure.

DETAILED DESCRIPTION:
Trabeculectomy is one of the most commonly performed glaucoma procedures performed to control IOP with approximately 18,000 operations performed in US Medicare beneficiaries alone in 2012. One complication of trabeculectomy surgery is the formation of subconjunctival and episcleral fibrosis, which occurs as part of the wound healing process and can result in fibrosis of the filtering bleb and failure. Transconjunctival needle revision (TCNR) aims to lyse subconjunctival adhesions and reestablish adequate aqueous humor flow from the anterior chamber to the subconjunctival space. One study reported 17% of trabeculectomies require bleb-needling revision. During TCNR the surgeon is able to visualize the trajectory of the needle or blade under the conjunctiva; however, detection of the fibrotic tissue and determination as to whether that tissue has been adequately lysed is difficult, limiting the success rate of the procedure.

Anterior segment optical coherence tomography (AS-OCT) allows for detailed assessment of the internal morphology of the bleb. Studies have utilized AS-OCT to assess morphological features of the bleb and correlate it with surgical success. A small case series reported the utility of AS-OCT for pre-operative planning for bleb revision, in particular, identifying safe access sites and minimizing conjunctival dissection.

More recently, real time OCT integrated with operative microscope has become available. Intraoperative OCT (iOCT) has been utilized extensively in retinal surgery and corneal surgery. Dada et al., described performing iOCT-guided TCNR in 2 patients with failed trabeculectomy blebs without intraoperative or postoperative complications. Investigators reported they were able to obtain a detailed view of the bleb wall and assess the depth and location of the needle, which permitted better lysis of adhesions. A pilot study by Kumar et al., reported one case of TCNR in which iOCT was used to demonstrate the extent of adhesions and loculations inside the bleb at the beginning of the procedure, and the lysis of these adhesions and formation of large single hyporeflective cavity inside the bleb at the end of the procedure. These small case studies suggest a role of iOCT imaging for TCNR, however, further research is needed to assess its feasibility and utility for routine use.

The aim of the research is to assess the surgical success, feasibility and utility of pre-operative Anterior Segment Optical Coherence Tomography (AS-OCT) and intraoperative Optical Coherence Tomography (iOCT) in trans-conjunctival needle revision (TCNR) of trabeculectomy bleb. Furthermore, investigators want to assess whether AS-OCT can be used to identify characteristics of trabeculectomy blebs that are associated with successful surgical outcomes.

To undergo this study, investigators will conduct a prospective study of patients who consent to AS-OCT and iOCT revision of TCNR. Investigators will compare the outcomes of these patients with retrospectively identified, historical controls (i.e. patients who underwent TCNR by the same surgeon without AS-OCT or iOCT assistance).

investigators hypothesize that information gained from pre-operative AS-OCT and intraoperative OCT will aid with intraoperative decision-making for TCNR of trabeculectomy bleb and will thereby improve surgical outcomes. Investigators also hypothesize that preoperative AS-OCT can be used to identify features of trabeculectomy bleb that can predict success with iOCT-assisted TCNR. More specifically, investigators hypothesize that filtering blebs with more extensive scarring as seen on pre-operative AS-OCT will benefit from iOCT.

ELIGIBILITY:
Inclusion criteria

* Briefly, the diagnosis of glaucoma is based on the presence of 2 or more of the following findings: 1) glaucomatous optic disc damage, defined as the presence of optic disc excavation, diffuse or focal neuroretinal rim thinning or notching, localized or generalized retinal nerve fiber layer (RNFL) thinning; 2) visual field defects consistent with glaucoma; and 3) IOP ≥ 22 mmHg.
* Patients with glaucoma who have been advised to undergo TCNR of a failed trabeculectomy bleb by a glaucoma specialist at Northwestern Medicine
* History of failed trabeculectomy (based on clinical features of the trabeculectomy bleb and elevated intraocular pressure)
* Patients can have history of other glaucoma surgery or cataract surgery
* The diagnosis of glaucoma is based on the presence of 2 or more of the following findings: 1) glaucomatous optic disc damage, defined as the presence of optic disc excavation, diffuse or focal neuroretinal rim thinning or notching, localized or generalized RNFL thinning; 2) visual field defects consistent with glaucoma; and 3) IOP ≥ 22 mmHg.

Exclusion criteria

* Age younger than 18 years;
* Secondary causes of glaucoma (e.g., iridocyclitis, trauma);
* Any evidence of corneal or conjunctival pathology adjacent to filtration bleb that could influence AS-OCT image
* Patients who did not undergo surgery or have adequate follow up
* Adults unable to consent, individuals who are not yet adults (infants, children, teenagers), pregnant women, prisoners and vulnerable populations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2022-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angelo P Tanna, MD, Principal Investigator — Professor
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arora KS, Robin AL, Corcoran KJ, Corcoran SL, Ramulu PY. Use of Various Glaucoma Surgeries and Procedures in Medicare Beneficiaries from 1994 to 2012. Ophthalmology. 2015 Aug;122(8):1615-24. doi: 10.1016/j.ophtha.2015.04.015. Epub 2015 Jun 16. PMID 26092196
- [Background] Kirwan JF, Lockwood AJ, Shah P, Macleod A, Broadway DC, King AJ, McNaught AI, Agrawal P; Trabeculectomy Outcomes Group Audit Study Group. Trabeculectomy in the 21st century: a multicenter analysis. Ophthalmology. 2013 Dec;120(12):2532-2539. doi: 10.1016/j.ophtha.2013.07.049. Epub 2013 Sep 23. PMID 24070811
- [Background] Mastropasqua R, Fasanella V, Agnifili L, Curcio C, Ciancaglini M, Mastropasqua L. Anterior segment optical coherence tomography imaging of conjunctival filtering blebs after glaucoma surgery. Biomed Res Int. 2014;2014:610623. doi: 10.1155/2014/610623. Epub 2014 Jul 20. PMID 25136603
- [Background] Hamanaka T, Omata T, Sekimoto S, Sugiyama T, Fujikoshi Y. Bleb analysis by using anterior segment optical coherence tomography in two different methods of trabeculectomy. Invest Ophthalmol Vis Sci. 2013 Oct 3;54(10):6536-41. doi: 10.1167/iovs.13-12439. PMID 23989189
- [Background] Kojima S, Inoue T, Kawaji T, Tanihara H. Filtration bleb revision guided by 3-dimensional anterior segment optical coherence tomography. J Glaucoma. 2014 Jun-Jul;23(5):312-5. doi: 10.1097/IJG.0b013e3182741ee6. PMID 23377583
- [Background] Ehlers JP, Modi YS, Pecen PE, Goshe J, Dupps WJ, Rachitskaya A, Sharma S, Yuan A, Singh R, Kaiser PK, Reese JL, Calabrise C, Watts A, Srivastava SK. The DISCOVER Study 3-Year Results: Feasibility and Usefulness of Microscope-Integrated Intraoperative OCT during Ophthalmic Surgery. Ophthalmology. 2018 Jul;125(7):1014-1027. doi: 10.1016/j.ophtha.2017.12.037. Epub 2018 Mar 2. PMID 29409662
- [Background] Dada T, Angmo D, Midha N, Sidhu T. Intraoperative Optical Coherence Tomography Guided Bleb Needling. J Ophthalmic Vis Res. 2016 Oct-Dec;11(4):452-454. doi: 10.4103/2008-322X.194150. PMID 27994819
- [Background] Kumar RS, Jariwala MU, V SA, Venugopal JP, Puttaiah NK, Balu R, Rao A S D, Shetty R. A Pilot Study on Feasibility and Effectiveness of Intraoperative Spectral-Domain Optical Coherence Tomography in Glaucoma Procedures. Transl Vis Sci Technol. 2015 Mar 9;4(2):2. doi: 10.1167/tvst.4.2.2. eCollection 2015 Mar. PMID 25767745
- [Background] Cantor LB, Mantravadi A, WuDunn D, Swamynathan K, Cortes A. Morphologic classification of filtering blebs after glaucoma filtration surgery: the Indiana Bleb Appearance Grading Scale. J Glaucoma. 2003 Jun;12(3):266-71. doi: 10.1097/00061198-200306000-00015. PMID 12782847

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: N/A. Single group, unmasked.
Units Other Than Participants: eyes
Groups:
- Study Group: Subjects scheduled to under trans-conjunctival needle revision
Period: Overall Study
Arm/Group | Study Group
Started | 10; 10 eyes
Completed | 7; 7 eyes
Not Completed | 3; 3 eyes
Not completed — Did not undergo surgery or did not undergo imaging at the time of surgery | 3

BASELINE CHARACTERISTICS:
Population: Subjects who underwent surgery and who underwent intra-operative imaging
Units Other Than Participants: Eyes
Groups:
- Study Group: Eyes scheduled to undergo trans-conjunctival needle revision of trabeculectomy bleb
Arm/Group | Study Group
Number analyzed (Participants) | 7
Number analyzed (Eyes) | 7
Age, Continuous [Mean (Full Range); unit: years] | 65.4 [51.5 to 80.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Number; unit: participants]
  United States | 7
Intraocular pressure (mmHg) [Mean (Full Range); unit: mm Hg] | 17.65 [12 to 22.5]

OUTCOME MEASURES:

1. Primary Outcome: Surgical Success
Description: Surgical success as defined as a 20% reduction in unmedicated IOP below the pre-operative baseline at specified post-operative visits.
Time Frame: Postoperative month 3
Population: Subjects who underwent trans-conjunctival needle revision and who underwent intra-operative imaging
Measure: Number; unit: participants
Units Other Than Participants: Eyes
Groups:
- Study Group: Subjects who underwent trans-conjunctival needle revision
Arm/Group | Study Group
Number analyzed (Participants) | 7
Number analyzed (Eyes) | 7
participants
  Success | 5
  Failure | 2

2. Secondary Outcome: Number of Participants With Successful Imaging of the Bleb With iOCT
Description: The secondary outcomes will be feasibility of intraoperative OCT. Feasibility will be defined as the percentage of cases with successful imaging of the bleb with iOCT.
Time Frame: Intraoperative assessment
Population: All eyes that underwent trans-conjunctival needle revision and intra-operative imaging
Measure: Number; unit: participants
Units Other Than Participants: Eyes
Arm/Group | Study Group
Number analyzed (Participants) | 7
Number analyzed (Eyes) | 7
participants | 7

3. Other Pre Specified Outcome: Pre-operative AS-OCT Findings
Description: Investigators will also assess whether findings seen with pre-operative AS-OCT can predict what type of blebs will benefit from iOCT-assisted TNCR. Features of AS-OCT and iOCT imaging that will be assessed include quality of image capture, visualization of surgical site, and characteristics of the bleb. Characteristics of the surgical site include bleb height, internal reflectivity, location and number of adhesions, and presence of cysts, cavities, and fistulas.
Time Frame: Pre-operative visit
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- Eyes Undergoing Trans-conjunctival Needle Revision: Open-angle glaucoma eyes that will undergo TCNR of trabeculectomy bleb
Arm/Group | Eyes Undergoing Trans-conjunctival Needle Revision
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2021-04-30): https://cdn.clinicaltrials.gov/large-docs/08/NCT05790408/Prot_002.pdf